CLINICAL TRIAL: NCT00260221
Title: Testing Interactions to Adjunctive Pain Control Techniques
Brief Title: VRH Pain Reduction During Burn Wound Care and Physical Therapy
Acronym: VRH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of General Medical Sciences (NIGMS) (NIH)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, David R. Patterson, PhD. ABPP. Professor, National Institute of General Medical Sciences (NIGMS)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19635-B; R01GM042725 (NIH)
Record Dates: First submitted 2005-11-30; First posted 2005-12-01 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2011-03

CONDITIONS: Burn
Keywords: Virtual Reality Hypnosis
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Arm one uses Virtual Reality Hypnosis post hypnotic suggestions to reduce pain durng wound care procedures.
  Interventions: Behavioral: using VR hypnosis/distraction and audio hypnosis
- 2 (Experimental): Arm two uses Virtual Reality distraction that is administered at times other than during burn care procedure to control for both for attention and high technology.
  Interventions: Behavioral: using VR hypnosis/distraction and audio hypnosis
- 3 (Experimental): Arm three use Audio administered Hypnosis without the visual technology.
  Interventions: Behavioral: using VR hypnosis/distraction and audio hypnosis

INTERVENTIONS:
Behavioral: using VR hypnosis/distraction and audio hypnosis — a between subject comparison using VR hypnosis and VR distraction and audio hypnosis for pain control

SUMMARY:
Using Virtual Reality Hypnosis to relief pain and anxiety for burn patients.

DETAILED DESCRIPTION:
The purpose of the study is to examine whether there is more effective relief of pain and anxiety during wound care procedures in burn-injured patients that are treated with Virtual Reality Hypnosis with post-hypnotic suggestion.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 7 years
* Able to complete subjective evaluations of pain
* English-speaking
* Not demonstrating delirium, psychosis, or any form of Organic Brain Disorder
* Able to communicate orally

Exclusion Criteria:

* Age less than 7 years
* Incapable of indicating subjective evaluation of pain
* Non-English-speaking
* Demonstrating delirium, psychosis, or Organic Brain Disorder
* Unable to communicate verbally
* Significant developmental disability
* Extreme susceptibility to motion sickness

Ages: 7 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2002-01; Primary Completion 2011-01 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
we use GRS, VAS, McGill,and nurse GRS to measure the pain. | once a day

CONTACTS AND LOCATIONS:
Overall Officials: David R. Patterson, Ph.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington; Harborview Medical Center, Seattle, Washington, United States

REFERENCES:
- [Background] Patterson DR, Tininenko JR, Schmidt AE, Sharar SR. Virtual reality hypnosis: a case report. Int J Clin Exp Hypn. 2004 Jan;52(1):27-38. doi: 10.1076/iceh.52.1.27.23925. PMID 14768967